CLINICAL TRIAL: NCT01566851
Title: Application of EULAR Recommendations for Cardiovascular Risk Management in Patients With Rheumatoid Arthritis in France in the Entire Population of the RSI (Other Branches of the Universal Healthcare Insurance Agency)
Brief Title: Application of EULAR Recommendations for Cardiovascular Risk Management in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 12-01
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Cardiovascular Check-up in Patients With Rheumatoid Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient: Patients with rheumatoid arthritis
  Interventions: Other: Cardiovascular check-up

INTERVENTIONS:
Other: Cardiovascular check-up — Cardiovascular check-up once a year in patients with rheumatoid arthritis

SUMMARY:
Introduction Cardiovascular diseases are the first cause of death in rheumatoid arthritis (RA). In 2010, EULAR Standing Committee for Clinical Affairs provides 10 recommendations for cardiovascular risk management in patients with rheumatoid arthritis, including a cardiovascular risk assessment annually.

The goal of this study is to evaluate the application of EULAR recommendations in real life in patients with RA in the french population. Inclusion criteria: all patients over 18 years old with rheumatoid arthritis treated with at least one DMARDS and/or biologic therapy, affiliated to the RSI (regime social des independents which correspond to other branches of the universal healthcare insurance agency). Non inclusion criteria: patients declared as rheumatoid arthritis without DMARDS or biologic therapy or treated with steroids alone. The following analysis will be performed on the whole database of the RSI, without name identification. Evaluation criteria: at least once a years the prescription of at least one of the following items use in the evaluation of the cardiovascular risk factors: lipides dosage, glycemia, HbA1C, stress test, Carotid ultra-sonography, coronary or lower limbs arteriography, heart ultra-sonography, cardiology clinic, endocrinology clinic. This evaluation will be done on the whole national population of RSI for the year 2011 (01/01/2011 - 31/12/2011). On a subgroup of patients from the region "Provence Alpes Côte d'Azur", the investigators will analyze the year 2009, and compare to year 2011, to evaluate the impact of theses recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, affiliated to RSI, with rheumatoid arthritis treated with at least one DMARDS and/or biologic therapy

Exclusion Criteria:

* patients under 18 years
* Patients declared as rheumatoid arthritis without DMARDS or biologic therapy or treated with steroids alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
the following items use in the evaluation of the cardiovascular risk factors | at time = 2 years
  At least once a years the prescription of at least one of the following items use in the evaluation of the cardiovascular risk factors:
  * Lipides dosage
  * Glycemia
  * HbA1C
  * Stress test
  * Carotid ultra-sonography
  * Coronary or lower limbs arteriography
  * Heart ultra-sonography
  * Cardiology clinic
  * Endocrinology clinic

SECONDARY OUTCOMES:
the following items use in the evaluation of the cardiovascular risk factors on the sub population | t=0 and t=2 years
  The same criteria of primary criteria but on the sub population of Povence Alpes Cote-d'Azur region a comparison of these criteria in 2009 (before EULAR recommendations ) and in 2011 (after EULAR recommendations)

CONTACTS AND LOCATIONS:
Overall Officials: Liana EULLER-ZIEGLER, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice